CLINICAL TRIAL: NCT05447494
Title: A Phase 1/2 Open-label, Dose Escalation Study Followed by a Multi-center, Randomized, Double-blind, Dose Comparison Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics of CAN103 in Newly Treated Gaucher Disease
Brief Title: Phase 1/2 Study of CAN103 in Subjects With Gaucher Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CANbridge (Suzhou) Bio-pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: CANbridge Life Sciences Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN103-GD-201; CTR20220507 (Registry Identifier: Center For Drug Evaluation, NMPA, China)
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Gaucher Disease, Type 1; Gaucher Disease, Type 3
Keywords: CAN103; Gaucher disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 is blinded to dose group. Except for the non-blind team, no other participants associated with this study should attempt to learn the treatment group assignment or which study treatment they are receiving. The unblinding of all subjects will take place after database lock.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose CAN103 (Experimental): Low dose intravenous infusion of CAN103 every other week for 37 weeks
  Interventions: Drug: Low-dose CAN103
- High-dose CAN103 (Experimental): High dose intravenous infusion of CAN103 every other week for 37 weeks
  Interventions: Drug: High-dose CAN103

INTERVENTIONS:
Drug: Low-dose CAN103 — Phase 1 is a within-subject dose escalation study to evaluate the safety, tolerability, and pharmacokinetics of two doses of CAN103 in newly treated subjects with GD1.
  Phase 2 is a randomized, double-blind, parallel group, dose comparison study to evaluate the efficacy and safety of two doses of CAN103 administered intravenously every other week for 37 weeks in newly treated GD1 or GD3 subjects with significant non-neurological clinical manifestations.
  Arms: Low-dose CAN103
Drug: High-dose CAN103 — Phase 1 is a within-subject dose escalation study to evaluate the safety, tolerability, and pharmacokinetics of two doses of CAN103 in newly treated subjects with GD1.
  Phase 2 is a randomized, double-blind, parallel group, dose comparison study to evaluate the efficacy and safety of two doses of CAN103 administered intravenously every other week for 37 weeks in newly treated GD1 or GD3 subjects with significant non-neurological clinical manifestations.
  Arms: High-dose CAN103

SUMMARY:
Gaucher disease is a rare lysosomal storage disorder caused by deficient activity of the enzyme acid β-glucosidase, causing glucosylceramide to accumulate within macrophages and leading to hepatosplenomegaly, anemia, thrombocytopenia, and bone disease. In the non-neuronpathic form (type 1), disease manifestations are mostly systemic, whereas in the neuronopathic forms, glucosylceramide also accumulates in the central nervous sysem and leads to acute (type 2) or chronic (type 3) neurodegeneration. The purpose of this Phase 1/2 first-in-human study is to initially evaluate the safety and tolerability of two doses of CAN103, and then barring any safety concerns, to evaluate the efficacy and safety of the two doses administered intravenously every other week in treatment-naive subjects with Gaucher disease type 1 or type 3.

DETAILED DESCRIPTION:
Phase 1: 4 newly treated subjects with Type I Gaucher disease (GD1). Phase 2: 36 newly treated subjects with GD1 or Type III Gaucher disease (GD3)

ELIGIBILITY:
Inclusion Criteria:

* Subjects have a confirmed clinical, enzymatic, and genetic diagnosis of Gaucher disease (Type 1 or Type 3);
* Phase 1: Subjects with GD1 aged ≥18 years; Phase 2: Subjects with GD1 or GD3 aged ≥12 years;
* Subjects have not received enzyme replacement therapy (ERT) or substrate replacement therapy (SRT) within 3 months before screening;
* Subjects have GD-related anemia and one or more of the following disease manifestations:

  1. Spleen volume ≥2 MN as measured by MRI, or
  2. Liver volume ≥1.5 MN as measured by MRI, or
  3. Platelet count ≥20 × 10^9/L and <100×10^9/L.

Exclusion Criteria:

* Subjects have received or stopped treatment with other investigational drugs or devices within 30 days before screening or less than 5 half-lives, whichever is longer (drugs only);
* Subjects have anemia due to other causes during screening, including nutritional anemia. Subjects whose nutritional anemia recovers with the treatment of iron, folic acid, or Vitamin B12 may be rescreened;
* Subjects have received hepatectomy or splenectomy;
* Subjects have had an allergic reaction to imiglucerase or other ERTs and their components;
* Subjects have received treatment with erythropoietin, whole blood or packed red blood cell transfusions, or chronic systemic corticosteroids within 3 months before screening, or have received a platelet transfusion within 1 month before screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in hemoglobin level from Baseline to Week 39 in the high-dose group | Baseline to Week 39
  Hemoglobin is measured in a central laboratory. An increase from Baseline indicates a therapeutic response.

SECONDARY OUTCOMES:
Mean percent change in platelet count from Baseline to Week 39 in the low-dose and high-dose groups. | Baseline to Week 39
  Platelet count is measured in a central laboratory. An increase in platelet count indicates a therapeutic response.
Mean percent change in liver volume (multiples of normal, MN) measured by magnetic resonance imaging (MRI) from Baseline to Week 39 in the low-dose and high-dose groups. | Baseline to Week 39
  Quantitative liver volume is calculated centrally by blinded radiologists. Normal liver volume is defined as 2.5% of body weight. A decrease from Baseline indicates a therapeutic response.
Mean percent change in spleen volume (MN) measured by MRI from Baseline to Week 39 in the low-dose and high-dose groups. | Baseline to Week 39
  Quantitative spleen volume is calculated centrally by blinded radiologists. Normal spleen volume is defined at 0.2% of body weight. A decrease in spleen volume indicates a therapeutic response.
Mean change in hemoglobin level from Baseline to Week 39 in the low-dose group. | Baseline and Week 39
  Hemoglobin is measured by a central laboratory. An increase from Baseline indicates a therapeutic response.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China